CLINICAL TRIAL: NCT05098444
Title: Endometriosis - Internet-based Therapy (Ed.iTh): Evaluation of an Internet-based Cognitive Behavioral Treatment to Improve the Quality of Life With Endometriosis
Brief Title: Efficacy of Internet-based Cognitive Behavioral Therapy for Endometriosis
Acronym: EdiTh
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Cornelia Weise, Dr. rer. nat., Philipps University Marburg
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CBT for endometriosis_2021
Record Dates: First submitted 2021-08-16; First posted 2021-10-28 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Endometriosis
Keywords: Endometriosis; Behavioral medicine; Internet based therapy; Cognitive behavioral therapy; Women's Health
MeSH Terms: conditions — Endometriosis | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Wait list control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral psychotherapy (Experimental): Internet-based CBT for patients with endometriosis:
  The experimental group has access to an online training consisting of 8 modules, one per week.
  Modules comprise of 1) psychoeducation (e.g., information about endometriosis and its treatment); 2) & 3) cognitive strategies (e.g., identifying and modifying dysfunctional cognitions); 4&5) pain and stress management (e.g. activity plans, relaxation techniques); 6) emotion regulation strategies (e.g. recognition and acceptance of emotions); 7) communication training (e.g. detection and communication of needs); 8) prophylaxis (e.g. summary of intervention, plans for the future).
  Participants are in weekly written contact with their assigned therapist via the news function of the training platform, receiving feedback on the content or getting answers to open questions.
  Interventions: Behavioral: Cognitive behavioral psychotherapy
- Waiting list (Other): During the waiting period, patients receive no treatment. After a waiting time of 5 months, patients of the waitlist receive the same iCBT treatment as the experimental group.
  Interventions: Other: Waiting list

INTERVENTIONS:
Behavioral: Cognitive behavioral psychotherapy — Internet-based Cognitive Behavioural Therapy aims to reduce the impairment due to endometriosis by using cognitive behavioural intervention techniques. Furthermore, therapy should enable the patients in coping with symptoms in the future.
  Arms: Cognitive behavioral psychotherapy
Other: Waiting list — Participants of the waiting list receive no treatment for 5 months. Afterwards they receive the same treatment as the experimental group.
  Arms: Waiting list

SUMMARY:
The purpose of this study is to evaluate the efficacy of an internet-based cognitive behavioral therapy in reducing the impairment caused by endometriosis.

DETAILED DESCRIPTION:
Endometriosis is a chronic disease in which endometrium-like (uterine lining-like) cells settle outside the uterus in the abdomen (Dunselman et al., 2014). The Endometriose Vereinigung Deutschland reports that between eight and 15 percent of all women during reproductive age are affected and that there are 40,000 new cases annually in Germany (Endometriose Vereinigung Deutschland e.V., 2020). Thus, endometriosis is the second most common gynecological disease. Despite the high prevalence, the etiology and pathogenesis of many factors remains unclear. Misdiagnoses are common and to reach the correct diagnosis it takes an average of 5 to 8.9 years (Chaman-Ara, Bahrami & Bahrami, 2017). So far there is no curative treatment option and the primarily medical treatment options are sometimes associated with serious side effects (Moradi, Parker, Sneddon, Lopez & Ellwood, 2014). Endometriosis is characterized by a multitude of physical as well as considerable psychological symptoms that significantly reduce the quality of life of those affected (Gao et al., 2006). For example, endometriosis is associated with higher levels of depression and anxiety disorders (Pope, Sharma, Sharma & Mazmanian, 2015). A psychotherapeutic supplement to the primary medical treatment to promote disease coping and expansion of coping strategies therefore appears sensible.

In the planned study, a CBT program specifically for endometriosis sufferers will therefore be developed and evaluated.

Previous intervention studies aimed at improving the quality of life of endometriosis sufferers examined mind-body interventions such as yoga (Gonçalves, Barros & Bahamondes, 2017), relaxation training (Zhao et al., 2012) and acupuncture in combination with conversational psychotherapy (Meissner et al., 2016). Hansen et al. (2017) were able to show in an uncontrolled pilot study (N = 10) that mindfulness-based psychotherapy significantly reduces the burden of endometriosis. Overall, the number of psychological intervention studies on endometriosis is very low and their quality often requires a critical classification due to methodological limitations (for an overview see Evans, Fernandez, Olive, Payne & Mikocka-Walus, 2019; Van Niekerk, Weaver-Pirie & Matthewson, 2019). Numerous evidence of effectiveness from the area of chronic pain disorders (Williams, Fisher, Hearn & Eccleston, 2020) as well as disorders in the area of women's health such as premenstrual dysphoric disorder (PMDD, Weise et al., 2019) undermine a possible effectiveness of CBT in endometriosis. To the best of our knowledge, however, there is no study to date that has tested the effectiveness of CBT for improving the quality of life of endometriosis sufferers.

The treatment program developed as part of the planned study is to be implemented as an internet-based intervention. A large number of studies confirm the effectiveness of internet-based CBT (iCBT) in various mental (Loughnan, Joubert, Grierson, Andrews & Newby, 2019), psychosomatic (Andersson, Cuijpers, Carlbring, Riper & Hedman, 2014) and somatopsychic diseases (Bernardy, Füber, Köllner & Häuser, 2010). The iCBT has now established itself as being as effective as face-to-face therapy (Carlbring, Andersson, Cuijpers, Riper & Hedman-Lagerlöf, 2018; Andersson, Carlbring & Rozental, 2019)

The internet-based implementation in the present study has various advantages: On the one hand, the effectiveness of the iCBT can be checked efficiently and in a resource-saving manner (Hedman, Andersson, Ljoeétsson, Axelsson & Lekander, 2016). On the other hand, endometriosis sufferers can be addressed throughout the German-speaking area, which ensures that a sufficient sample size can be achieved. Ultimately, those affected that would otherwise not receive any treatment due to the lack of regional availability of interventions, also have access to treatment. In addition, issues such as the desire to have children and endometriosis often lead to shame. An intervention offered online and anonymously can encourage the use of assistance here.

The aim of the study is to examine the effectiveness of iCBT in reducing the stress and impairment caused by endometriosis and in increasing the health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* People with female-assigned reproductive systems aged 18 to 45 years
* Medically confirmed endometriosis diagnosis
* Impairment of quality of life due to endometriosis defined as a value of ≥ 15 points across all scales in the Endometriosis Health Profile 30 + 23 (EHP-30 + 23, (Jones, Kennedy, Barnard, Wong & Jenkinson, 2001a)
* Adequate German language skills
* Access to a personal computer (PC) / laptop and adequate internet connection

Exclusion Criteria:

* Serious mental disorder: unipolar severe depression (Beck Depression Inventory II: raw value ≥ 29), presuicidal syndrome, bipolar affective disorder, unipolar mania, psychotic disorder, alcohol or substance dependence
* Psychotherapeutic treatment: currently or within the last two years
* Use of benzodiazepines (prevents learning processes that are important for psychotherapy)
* Changes in the intake or use (e.g. start / change of dose / discontinuation) of antidepressants and hormonal contraceptives within the last three months
* Current or planned intrauterine insemination (IUI), in-vitro-fertilisation (IVF) or intracytoplasmic sperm injection (ICSI) treatment with hormonal stimulation within the next eight months
* Suffering from one of the following diseases: malignant tumor, in particular breast, cervical or ovarian cancer, ulcerative colitis, Crohn's disease, a known bacterial or viral infection (e.g. tuberculosis (TBC), hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV)
* Current pregnancy or birth of a child within the last six months, breastfeeding within the last six months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Endometriosis Health Profile 30 + 23 (EHP-30 + 23; Jones, Kennedy, Barnard, Wong & Jenkinson, 2001) | Pre-treatment (baseline), post-treatment (change from basline at 8-10 weeks after treatment start), change from baseline 3 month after treatment start, change from baseline 12 month after treatment start
  Assessment of impairment of endometriosis-related quality of life (long version)(self-rating)
Change in Endometriosis Health Profile 5 (EHP-5; Jones, Jenkinson & Kennedy, 2004) | Pre-treatment (baseline), change from baseline weekly during treatment, change from basline at 8-10 weeks after treatment start, change from baseline 3 month after treatment start, change from baseline 12 month after treatment start
  Assessment of impairment of endometriosis-related quality of life (short version)(self-rating)
Change in Pain Disability Index (PDI; Tait, Pollard & Margolis, 1987) | Pre-treatment (baseline), post-treatment (change from basline at 8-10 weeks after treatment start), change from baseline 3 month after treatment start, change from baseline 12 month after treatment start
  Assessment of impairment due to pain (self-rating)
Change in Visual analog pain scale (VAS) | Pre-treatment (baseline), change from baseline weekly during treatment, change from basline at 8-10 weeks after treatment start, change from baseline 3 month after treatment start, change from baseline 12 month after treatment start
  Assessment of impairment due to pain during menstruation and at the moment (self-rating)

SECONDARY OUTCOMES:
Change in Brief Patient Health Questionnaire (PHQ-9; Zipfel, Herzog & Löwe, 2004) | Pre-treatment (baseline), post-treatment (change from basline at 8-10 weeks after treatment start), change from baseline 3 month after treatment start, change from baseline 12 month after treatment start
  Assessment of depressive mood (self-rating)
Change in Perceived Stress Scale (PSS; Klein et al., 2016) | Pre-treatment (baseline), post-treatment (change from basline at 8-10 weeks after treatment start), change from baseline 3 month after treatment start, change from baseline 12 month after treatment start
  Assessment of perceived stress (self-rating)
Change in Brief Cope (Carver, 1997) | Pre-treatment (baseline), post-treatment (change from basline at 8-10 weeks after treatment start), change from baseline 3 month after treatment start, change from baseline 12 month after treatment start
  Assessment of coping skills (self-rating)
Change in Illness Perception Questionnaire (IPQ-R; Glattacker, Bengel & Jäckel, 2009) | Pre-treatment (baseline), post-treatment (change from basline at 8-10 weeks after treatment start), change from baseline 3 month after treatment start, change from baseline 12 month after treatment start
  Assessment of cognitive representation of illness (self-rating)
Change in The Acceptance and Action Questionnaire - II (FAH-II; Hoyer & Gloster, 2013) | Pre-treatment (baseline), post-treatment (change from basline at 8-10 weeks after treatment start), change from baseline 3 month after treatment start, change from baseline 12 month after treatment start
  Assessment of psychological flexibility (self-rating)

OTHER OUTCOMES:
Relationship Assessment Scale (RAS; Hendrick, 1988) | Pre-treatment
  Assessment of quality of partnership (self-rating)
Big Five Inventory - 10 (BFI-10; Rammstedt & John, 2007) | Pre-treatment
  Assessment of personality factors (self-rating)
Negative Effects of Psychological Treatment Questionnaire (NEQ; Rozental, Kottorp, Boettcher & Andersson, 2016) | Post-treatment (8-10 weeks after treatment start), 3-month-follow-up, 12-month-follow-up
  Assessment of side effects of the intervention (self-rating)
Satisfaction with treatment (self developed questionnaire) | Weekly during treatment, post-treatment (8-10 weeks after treatment start), 3-month-follow-up, 12-month-follow-up
  Assessment of satisfaction with treatment (self-rating)
Web-Based Screening Questionnaire (WSQ, Donker, Van Straten, Marks & Cuijpers, 2009) | Screening (up to 4 weeks before treatment start)
  Assessment of inclusion and exclusion criteria
International Diagnosis Checklist for International Classification of Diseases (ICD-10) (IDCL; Hiller et al., 2004) | Screening (up to 4 weeks before treatment start)
  Telephone interview, assessment of inclusion and exclusion criteria

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Weise, Ph.D, Principal Investigator — Philipps University Marburg
Locations (1):
- Philipps University Marburg, Dept. of Psychology, Division of Clinical Psychology and Psychotherapy, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Depends on the sample size. Patient data are highly sensible and anonymization might be threatened if the sample size is too small.

REFERENCES:
- [Background] Klein EM, Brahler E, Dreier M, Reinecke L, Muller KW, Schmutzer G, Wolfling K, Beutel ME. The German version of the Perceived Stress Scale - psychometric characteristics in a representative German community sample. BMC Psychiatry. 2016 May 23;16:159. doi: 10.1186/s12888-016-0875-9. PMID 27216151
- [Background] Jones G, Kennedy S, Barnard A, Wong J, Jenkinson C. Development of an endometriosis quality-of-life instrument: The Endometriosis Health Profile-30. Obstet Gynecol. 2001 Aug;98(2):258-64. doi: 10.1016/s0029-7844(01)01433-8. PMID 11506842
- [Background] Jones G, Jenkinson C, Kennedy S. Development of the Short Form Endometriosis Health Profile Questionnaire: the EHP-5. Qual Life Res. 2004 Apr;13(3):695-704. doi: 10.1023/B:QURE.0000021321.48041.0e. PMID 15130031
- [Background] Hoyer, J. & Gloster, A. T. (2013). Fragebögen und Skalen · Questionnaires and Scales Verhaltenstherapie 2013;23:42-44 Psychologische Flexibilität messen: Der Fragebogen zu Akzeptanz und Handeln II. https://doi.org/10.1159/000347040
- [Background] Hendrick, S. S. (1988). A Generic Measure of Relationship Satisfaction. Journal of Marriage and the Family, 50(1), 93. https://doi.org/10.2307/352430
- [Background] Hiller, W., Zaudig, M. & Mombour, W. (2004). IDCL-Internationale Diagnosen Checklisten für DSM-IV und ICD-10 [Inter-national Diagnostic Checklists for DSM-IV and ICD-10] (Band 2). Bern: Huber.
- [Background] Hahlweg, K. (1979). Konstruktion und Validierung des Partnerschaftsfragebogen PFB. Zeitschrift für Klinische Psychologie, 8(1).
- [Background] Glattacker, M., Bengel, J. & Jäckel, W. H. (2009). Die deutschsprachige Version des Illness Perception Questionnaire-revised: Psychometrische Evaluation an Patienten mit chronisch somatischen Erkrankungen. Zeitschrift fur Gesundheitspsychologie, 17(4), 158-169. Hogrefe Verlag Göttingen . https://doi.org/10.1026/0943-8149.17.4.158
- [Background] Donker T, van Straten A, Marks I, Cuijpers P. A brief Web-based screening questionnaire for common mental disorders: development and validation. J Med Internet Res. 2009 Jul 24;11(3):e19. doi: 10.2196/jmir.1134. PMID 19632977
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Rammstedt, B. & John, O. P. (2007). Measuring personality in one minute or less: A 10-item short version of the Big Five Inventory in English and German. Journal of Research in Personality, 41, 203-212. https://doi.org/10.1016/j.jrp.2006.02.001
- [Background] Rozental A, Kottorp A, Boettcher J, Andersson G, Carlbring P. Negative Effects of Psychological Treatments: An Exploratory Factor Analysis of the Negative Effects Questionnaire for Monitoring and Reporting Adverse and Unwanted Events. PLoS One. 2016 Jun 22;11(6):e0157503. doi: 10.1371/journal.pone.0157503. eCollection 2016. PMID 27331907
- [Background] Tait RC, Pollard CA, Margolis RB, Duckro PN, Krause SJ. The Pain Disability Index: psychometric and validity data. Arch Phys Med Rehabil. 1987 Jul;68(7):438-41. PMID 3606368
- [Background] Zipfel, S., Herzog, W. & Löwe, B. (2004). Screening psychischer Störungen mit dem "Gesundheitsfragebogen für Patienten (PHQ-D)". Diagnostica, 50(4), 171-181. https://doi.org/10.1026/0012-1924.50.4.171
- [Background] Endometriose Vereinigung Deutschland e.V. (2020). Was ist Endometriose? Zugriff am 21.12.2020. Verfügbar unter: https://www.endometriose-vereinigung.de/was-ist-endometriose.html
- [Result] Dunselman GA, Vermeulen N, Becker C, Calhaz-Jorge C, D'Hooghe T, De Bie B, Heikinheimo O, Horne AW, Kiesel L, Nap A, Prentice A, Saridogan E, Soriano D, Nelen W; European Society of Human Reproduction and Embryology. ESHRE guideline: management of women with endometriosis. Hum Reprod. 2014 Mar;29(3):400-12. doi: 10.1093/humrep/det457. Epub 2014 Jan 15. PMID 24435778
- [Result] Chaman-Ara, K., Bahrami, M. A. & Bahrami, E. (2017). Endometriosis psychological aspects: A literature review. Journal of Endometriosis and Pelvic Pain Disorders, 9(2), 105-111. https://doi.org/10.5301/jeppd.5000276
- [Result] Moradi M, Parker M, Sneddon A, Lopez V, Ellwood D. Impact of endometriosis on women's lives: a qualitative study. BMC Womens Health. 2014 Oct 4;14:123. doi: 10.1186/1472-6874-14-123. PMID 25280500
- [Result] Gao X, Yeh YC, Outley J, Simon J, Botteman M, Spalding J. Health-related quality of life burden of women with endometriosis: a literature review. Curr Med Res Opin. 2006 Sep;22(9):1787-97. doi: 10.1185/030079906X121084. PMID 16968582
- [Result] Pope CJ, Sharma V, Sharma S, Mazmanian D. A Systematic Review of the Association Between Psychiatric Disturbances and Endometriosis. J Obstet Gynaecol Can. 2015 Nov;37(11):1006-15. doi: 10.1016/s1701-2163(16)30050-0. PMID 26629721
- [Result] Goncalves AV, Barros NF, Bahamondes L. The Practice of Hatha Yoga for the Treatment of Pain Associated with Endometriosis. J Altern Complement Med. 2017 Jan;23(1):45-52. doi: 10.1089/acm.2015.0343. Epub 2016 Nov 21. PMID 27869485
- [Result] Zhao L, Wu H, Zhou X, Wang Q, Zhu W, Chen J. Effects of progressive muscular relaxation training on anxiety, depression and quality of life of endometriosis patients under gonadotrophin-releasing hormone agonist therapy. Eur J Obstet Gynecol Reprod Biol. 2012 Jun;162(2):211-5. doi: 10.1016/j.ejogrb.2012.02.029. Epub 2012 Mar 26. PMID 22455972
- [Result] Meissner K, Schweizer-Arau A, Limmer A, Preibisch C, Popovici RM, Lange I, de Oriol B, Beissner F. Psychotherapy With Somatosensory Stimulation for Endometriosis-Associated Pain: A Randomized Controlled Trial. Obstet Gynecol. 2016 Nov;128(5):1134-1142. doi: 10.1097/AOG.0000000000001691. PMID 27741200
- [Result] Hansen, K. E., Kesmodel, U. S., Kold, M. & Forman, A. (2017). Long-term effects of mindfulness-based psychological intervention for coping with pain in endometriosis: A six-year follow-up on a pilot study. Nordic Psychology, 69(2), 100-109. Routledge. https://doi.org/10.1080/19012276.2016.1181562
- [Result] Evans S, Fernandez S, Olive L, Payne LA, Mikocka-Walus A. Psychological and mind-body interventions for endometriosis: A systematic review. J Psychosom Res. 2019 Sep;124:109756. doi: 10.1016/j.jpsychores.2019.109756. Epub 2019 Jun 27. PMID 31443810
- [Result] Van Niekerk L, Weaver-Pirie B, Matthewson M. Psychological interventions for endometriosis-related symptoms: a systematic review with narrative data synthesis. Arch Womens Ment Health. 2019 Dec;22(6):723-735. doi: 10.1007/s00737-019-00972-6. Epub 2019 May 12. PMID 31081520
- [Result] Williams ACC, Fisher E, Hearn L, Eccleston C. Psychological therapies for the management of chronic pain (excluding headache) in adults. Cochrane Database Syst Rev. 2020 Aug 12;8(8):CD007407. doi: 10.1002/14651858.CD007407.pub4. PMID 32794606
- [Result] Weise C, Kaiser G, Janda C, Kues JN, Andersson G, Strahler J, Kleinstauber M. Internet-Based Cognitive-Behavioural Intervention for Women with Premenstrual Dysphoric Disorder: A Randomized Controlled Trial. Psychother Psychosom. 2019;88(1):16-29. doi: 10.1159/000496237. Epub 2019 Feb 19. PMID 30783069
- [Result] Loughnan SA, Joubert AE, Grierson A, Andrews G, Newby JM. Internet-delivered psychological interventions for clinical anxiety and depression in perinatal women: a systematic review and meta-analysis. Arch Womens Ment Health. 2019 Dec;22(6):737-750. doi: 10.1007/s00737-019-00961-9. Epub 2019 May 17. PMID 31101993
- [Result] Andersson G, Cuijpers P, Carlbring P, Riper H, Hedman E. Guided Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: a systematic review and meta-analysis. World Psychiatry. 2014 Oct;13(3):288-95. doi: 10.1002/wps.20151. PMID 25273302
- [Result] Bernardy K, Fuber N, Kollner V, Hauser W. Efficacy of cognitive-behavioral therapies in fibromyalgia syndrome - a systematic review and metaanalysis of randomized controlled trials. J Rheumatol. 2010 Oct;37(10):1991-2005. doi: 10.3899/jrheum.100104. Epub 2010 Aug 3. PMID 20682676
- [Result] Andersson G, Carlbring P, Rozental A. Response and Remission Rates in Internet-Based Cognitive Behavior Therapy: An Individual Patient Data Meta-Analysis. Front Psychiatry. 2019 Oct 25;10:749. doi: 10.3389/fpsyt.2019.00749. eCollection 2019. PMID 31708813
- [Result] Carlbring P, Andersson G, Cuijpers P, Riper H, Hedman-Lagerlof E. Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: an updated systematic review and meta-analysis. Cogn Behav Ther. 2018 Jan;47(1):1-18. doi: 10.1080/16506073.2017.1401115. Epub 2017 Dec 7. PMID 29215315
- [Result] Hedman E, Andersson E, Ljotsson B, Axelsson E, Lekander M. Cost effectiveness of internet-based cognitive behaviour therapy and behavioural stress management for severe health anxiety. BMJ Open. 2016 Apr 25;6(4):e009327. doi: 10.1136/bmjopen-2015-009327. PMID 27113231
- [Derived] Schubert K, Lohse J, Kalder M, Ziller V, Weise C. Internet-based cognitive behavioral therapy for improving health-related quality of life in patients with endometriosis: study protocol for a randomized controlled trial. Trials. 2022 Apr 12;23(1):300. doi: 10.1186/s13063-022-06204-0. PMID 35414092